CLINICAL TRIAL: NCT05026957
Title: A Shared Decision Making Approach With Digital Support to Improve Quality of Life, Exercise Capacity, Motivation to Exercise, Perception of Rehabilitation and Engagement in the Decision Making Process in Patients With Coronary Artery Disease in a Cardiac Rehabilitation Setting
Brief Title: A Digitally-Supported Shared Decision Making Approach for Coronary Artery Disease Patients During Cardiac Rehabilitation
Acronym: SharedHeart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, Head of Cardiology, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19.09/cardio 19.03
Record Dates: First submitted 2021-08-12; First posted 2021-08-30 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Cardiac Rehabilitation; Digital Health; Telerehabilitation

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participating in regular cardiac rehabilitation
  Interventions: Device: SharedHeart
- Intervention (Experimental): Participating in regular cardiac rehabilitation + using the shared-decision making application
  Interventions: Device: SharedHeart

INTERVENTIONS:
Device: SharedHeart — A smartphone application

SUMMARY:
Investigating the role of shared-decision making in cardiac rehabilitation

DETAILED DESCRIPTION:
The clinical study is a prospective double-arm, randomized controlled trial to study the user experience of the approach with the supporting applications, and the impact on patients' quality of life, physical activity, perception of rehabilitation and engagement in the decision making process.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of coronary artery disease with or without intervention (PCI/CABG/conservative)
* Be clinically stable without inducible ischemia or high risk ventricular arrhythmia, confirmed by the last available maximal ergospirometry test
* Recently having started cardiac rehabilitation in Jessa Hospital Hasselt
* Age ≥18 years
* Willing and physically able to follow a technology-supported shared decision making program and other study procedures in a three months follow-up period
* Show evidence of a personally signed and dated informed consent, indicating that the subject (or a legally-recognized representative) has been informed of all pertinent aspects of the study
* Possession of and/or able to use an Android based smartphone
* Possession of internet connectivity
* Dutch speaking and understanding

Exclusion Criteria:

* • Orthopedic, neurologic or any other pathologic condition which makes the patient physically unable to follow a technology-supported shared decision making program

  * Planned interventional procedure or surgery in the next three months
  * Pregnant females
  * Present cardiovascular complaints
  * Participation in other cardiac rehabilitation program trials, focusing on exercise outcome
  * Current or recent participation in other technology-supported programs, even when not directly targeting exercise capacity
  * Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study or a life expectancy of less than three months based on investigators judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart-related Quality of Life | 3 months
  The Heart-related Quality of Life will be assesed with a validated questionnaire "HeartQoL". The questionnaire will be administered to the patient at baseline and after 3 months on paper.

SECONDARY OUTCOMES:
Exercise capacity change | 3 months
  Peak VO2 with CPET

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No